CLINICAL TRIAL: NCT05205096
Title: Study on the Immunogenicity and Safety of Booster Immunization of Recombinant Novel Coronavirus Vaccine (CHO Cells) After Inoculation With Two Doses of Inactivated Vaccine (CoronaVac) in People Over 18 Years Old
Brief Title: Immunogenicity and Safety of Booster Immunization of ZF2001 After Inoculation With Two Doses of CoronaVac
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT-LKM-2021-NCV03-02
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational vaccine group (Experimental): Recombinant novel coronavirus vaccine (CHO cells) injection, Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose.
  Interventions: Biological: Recombinant novel coronavirus vaccine (CHO cells)

INTERVENTIONS:
Biological: Recombinant novel coronavirus vaccine (CHO cells) — At 3-9 months after the immunization with 2 doses of inactivated vaccine (CoronaVac), 1 dose of recombinant novel coronavirus vaccine (CHO cells) is vaccinated.

SUMMARY:
Study objectives: To evaluate the immunogenicity and immunity persistence and safety of recombinant novel coronavirus vaccine (CHO cells) after booster immunization in populations vaccinated with two doses of marketed novel coronavirus inactivated vaccine (CoronaVac).

Study method: For the subjects who have been vaccinated with two doses (the interval between two doses ≥ 3 weeks) of the novel coronavirus inactivated vaccine (CoronaVac) for 3 to 9 months, 1 dose of the recombinant novel coronavirus vaccine (CHO cells) was administered. Blood samples were collected before booster immunization, 14 days, 30 days and 180 days after booster immunization for neutralizing antibody detection.

All AEs were collected within 1 month after the booster immunization. All SAEs were collected within 6 months after the booster immunization.

DETAILED DESCRIPTION:
This trial plans to enroll 480 subjects, who will be divided into 3 groups according to the interval between booster immunization and basic immunization: group A (3-4 months), group B (5-6 months), group C (7-9 months) each with 160 subjects (including 120 subjects aged 18-59 years and 40 subjects aged 60 years and above).

The recombinant novel coronavirus vaccine (CHO cells) was thoroughly mixed and injected intramuscularly at the deltoid muscle of the upper arm according to the instructions. Blood samples were collected before booster immunization, 14 days, 30 days and 180 days after booster immunization for neutralizing antibody detection.

All AEs were collected within 1 month after the booster immunization. Solicited AEs (the following events occurring within 7 days of vaccination) :

Adverse events at the inoculation site (local) : pain, pruritus, redness, swelling, rash, induration; Non-inoculated site (systemic) adverse events: fever, headache, fatigue, diarrhea, nausea, vomiting, muscle pain (non-inoculated site), acute allergic reactions, cough.

All SAEs were collected within 6 months after the booster immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people over 18 years old, and can provide vaccination information to prove that they have completed 2 doses of inactivated novel coronavirus vaccine (CoronaVac) within the past 3-9 months;
* The subjects voluntarily participate in the research, sign the informed consent form, and can provide valid identification, understand and comply with the requirements of the study protocol;
* Female subjects of childbearing age agree to use effective contraception from the start of the study to 2 months after vaccination.

Exclusion Criteria:

* Suspected or confirmed fever (fever ≥38.5℃) within 72 hours before enrollment, or axillary body temperature ≥37.3℃ on the day of enrollment;
* Diastolic blood pressure ≥ 100 mmHg and/or systolic blood pressure ≥ 160 mmHg without or after drug control;
* Have a history of previous infection with new coronary pneumonia or a positive nucleic acid test history;
* Those who currently suffer from the following diseases: 1.Thrombocytopenia, any coagulation disorder, or receiving anticoagulant therapy, etc.; 2.History of congenital or acquired immunodeficiency or autoimmune disease; asplenia, or history of spleen surgery, trauma, or treatment with immunomodulatory agents within 6 months, such as: immunosuppressive doses of glucocorticoids (dose reference: equivalent or prednisone 20mg/day for more than one week); or monoclonal antibody; or thymosin; or interferon, etc.; 3.Those suffering from acute infectious diseases or using antipyretic/analgesic/antiallergic drugs within 3 days before enrollment, or acute exacerbation of chronic diseases; 4.Cancer patients (except basal cell carcinoma) who have been off treatment for less than 6 months; 5.Serious chronic diseases such as congenital heart disease, severe liver and kidney disease, severe diabetes (with complications) that may interfere with the conduct or completion of the study; 6.Active tuberculosis, viral hepatitis patients with obvious liver damage (excluding virus carriers) and/or HIV-positive or syphilis-specific antibody-positive;
* Previous history of severe hypersensitivity to any vaccine, or severe hypersensitivity history to any component of the investigational vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, dyspnea, vascular nerve edema, etc.;
* Administer subunit vaccine and inactivated vaccine within 14 days before the trial vaccine, and receive live attenuated vaccine within 28 days;
* Received blood or blood-related products, including immune globulin, within 3 months prior to screening; or planned use within 6 months after study initiation to full vaccination;
* In addition to completing 2 doses of inactivated novel coronavirus vaccine within the past 3-9 months, participating in other COVID-19 related clinical trials;
* Pregnant women (including women of childbearing age with positive urine pregnancy test);
* Investigators believe that the presence of any disease or condition in the subject may put the subject at unacceptable risk; the subject cannot meet protocol requirements; interfere with the assessment of vaccine response, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity endpoint | 14 days after booster vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody

SECONDARY OUTCOMES:
Immunogenicity endpoint | 30, 180 days after booster vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody
Immunogenicity endpoint | 14 days, 30 days, and 180 days after booster vaccination
  4 times growth rate of SARS-CoV-2 neutralizing antibody
Safety endpoint | Within 1 month after booster vaccination
  Incidence of AEs
Safety endpoint | Within 6 months after booster vaccination
  Incidence of SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Huakun Lv, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No